CLINICAL TRIAL: NCT05182385
Title: An Open Label, Phase I/II Study of Venetoclax in Addition to Blinatumomab Immunotherapy in Adult Patients With Relapsed/Refractory B Cell Precursor Acute Lymphoblastic Leukemia (BCP-ALL)
Brief Title: Venetoclax in Addition to Blinatumomab in Adult Patients With Relapsed/Refractory B Cell Precursor Acute Lymphoblastic Leukemia Relapsed/Refractory B Cell Precursor Acute Lymphoblastic Leukemia (BCP-ALL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Principal Investigator, Goethe University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL-BLIVEN; 2021-001384-25 (EudraCT Number)
Record Dates: First submitted 2021-12-17; First posted 2022-01-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: ALL, Recurrent, Adult
Keywords: ALL; acute lymphoblastic leukemia; MRD positive; minimal residual disease; blinatumomab; venetoclax
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hematological relapse (Experimental): Diagnosis of Ph-negative, CD19-positive B-precursor acute lymphoblastic leukemia according to WHO classification:
  * Refractory BCP-ALL to primary induction therapy, including at least three cycles of standard chemotherapy
  * Untreated first relapse of BCP-ALL with first remission duration < 12 months or
  * Second or greater relapse of BCP-ALL or refractory relapse or
  * Relapse of BCP-ALL any time after allogeneic HSCT
  Interventions: Drug: Blinatumomab; Drug: Venetoclax
- molecular relapse (Experimental): Diagnosis of Ph-negative, CD19-positive B-precursor acute lymphoblastic leukemia according to WHO classification:
  -Positivity of MRD marker of immunoglobulin/T-cell receptor gene rearrangements of greater than 0.01% if in first or second remission of BCP-ALL
  Interventions: Drug: Blinatumomab; Drug: Venetoclax

INTERVENTIONS:
Drug: Blinatumomab — All patients with hematological relapse will additionally receive Blinatumomab immunotherapy (first cycle: 9 ug/d c.i.v. on d1 until d7 and 28 ug/d c.iv. on d8 until d28; second cycle: 28 ug/d c.iv. on d1 to d28) in six-week cycles (4 weeks on Blinatumomab, 2 weeks off Blinatumomab).
  All patients with molecular relapse will additionally receive Blinatumomab immunotherapy at 28 ug/d c.iv. on d1 until d28 in six-week cycles (4 weeks on Blinatumomab, 2 weeks off Blinatumomab.)
  Patients eligible for a second cycle shall not receive Blinatumomab starting dose independent from relapse type.
  Other Names: blincyto
Drug: Venetoclax — In phase I of the study all eligible patients will receive increasing doses of Venetoclax on days -7 to -1 (Venetoclax dose-titration) in the first cycle and continuous dosing of Venetoclax at a pre-specified target dose (TD, p.o., once daily, d1 to d42) in six-week cycles for a maximum of two cycles.
  In phase II of the study all eligible patients will receive the recommended phase 2 dose (RP2D) of Venetoclax in six-week cycles for a maximum of two cycles. RP2D will be MTD.
  Patients eligible for a second cycle shall not receive Venetoclax dose-titration independent from relapse type.
  Other Names: Venclyxto

SUMMARY:
This study is designed to determine the feasibility, safety, tolerability and maximum tolerated dose of Venetoclax in combination with Blinatumomab and to evaluate the response in patients treated with the combination of Venetoclax and Blinatumomab in in patients with hematological relapse or molecular relapse.

DETAILED DESCRIPTION:
Transfer of patients to alloHSCT after one cycle or after a subsequent cycle is considered as per protocol discontinuation and as premature treatment discontinuation.

There will be a safety follow-up visit at 30 days after end of the last infusion. There will be efficacy follow-up until 6 months after end of therapy. In patients scheduled for SCT the 30-day safety-visit may be performed at the latest time point possible before initiation of subsequent treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
4. Availability of patient-specific molecular MRD markers of immunoglobulin/T-cell receptor gene rearrangementsas assessed by PCR with a sensitivity of at least 10E-04
5. Diagnosis of Philadelphia negative, CD19-positive B-precursor acute lymphoblastic leukemia according to WHO classification:

   * Refractory BCP-ALL to primary induction therapy, including at least three cycles of standard chemotherapy
   * Untreated first relapse of BCP-ALL with first remission duration < 12 months or
   * Second or greater relapse of BCP-ALL or refractory relapse or
   * Relapse of BCP-ALL any time after allogeneic HSCT or
6. Positivity of MRD marker of immunoglobulin/T-cell receptor gene rearrangements of greater than 0.01% if in first or second remission of BCP-ALL
7. Negative pregnancy test < 7 days before first study drug in women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they fulfil at least one of the following criteria:

   1. Post-menopausal (i.e. 12 months of natural amenorrhea or 6 months of amenorrhea with Serum FSH > 40 U/ml
   2. Post-operative after bilateral ovariectomy with or without hysterectomy
   3. Continuous and correct application of a contraception method with a Pearl index of < 1% (e.g. implants, depots, oral contraceptives, intrauterine device) from initial study drug administration until at least 3 months after the last dose of study drug. A hormonal contraception method must always be combined with a barrier method (e.g. condom)
   4. Sexual abstinence
   5. Vasectomy of the sexual partner
8. Ability to understand and willingness to sign a written informed consent
9. Willingness to participate in the registry of the German Multicenter Study Group for Adult ALL (GMALL)

Exclusion Criteria:

1. Patients with diagnosis of Philadelphia positive BCP-ALL according to WHO classifiation
2. Patients with diagnosis of Burkitt´s Leukemia according to WHO classification
3. Patients with extramedullary relapse; non-bulky lymph node (< 7.5 cm diameter) involvement will be accepted
4. Patients with CNS involvement at relapse (as determined by CSF analysis)
5. Patients with suspected or histologically confirmed testicular involvement at relapse
6. Current autoimmune disease of any kind or history of autoimmune disease with potential CNS involvement
7. Patients with Philadelphia-positive BCP-ALL still receiving TKI
8. Prior or concomitant therapy with BH3 mimetics
9. Prior therapy with anti CD19 therapy, unless administered in MRD-positive setting (i.e. with bone marrow blasts ≤ 5%)
10. Treatment with any of the following within 7 days prior to the first dose of study drug: strong cytochrome P450 3A (CYP3A) inhibitors, moderate or strong CYP3A inducers
11. Intake of any of the following within 3 days prior to the first dose of study drug: grapefruit, grapefruit products, Seville oranges or star fruit
12. Presence of Graft-versus-Host Disease (GvHD) and/or on immunosuppressant medication within 2 weeks before start of protocol-specified therapy
13. Radiation, chemotherapy (with the exception of prephase therapy), or immunotherapy or any other anticancer therapy ≤ 2 weeks prior to Cycle 1 Day 1 or radio-immunotherapy 4 weeks prior to Cycle 1 Day 1.
14. Major surgery within 2 weeks of first dose of study drug
15. Patients who are pregnant or lactating
16. Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety
17. Unstable cardiovascular function:

    * Symptomatic ischemia, or
    * Uncontrolled clinically significant conduction abnormalities (1st degree AV block or asymptomatic LAFB/RBBB will not be excluded), or
    * Congestive heart failure (CHF) of NYHA Class ≥3, or
    * Myocardial infarction (MI) within 3 months
18. Evidence of clinically significant uncontrolled condition(s) including, but not limited to: Uncontrolled and/or active systemic infection (viral, bacterial or fungal), chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti- HBs antibody (anti-HBs) positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) or blood transfusions may participate.
19. Known human immunodeficiency virus (HIV) infection (HIV testing is not required)
20. Patients unable to swallow tablets, patients with malabsorption syndrome, or any other GI disease or GI dysfunction that could interfere with absorption of study treatment
21. Adequate hepatic function per local laboratory reference range as follows: Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0X ULN, Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
22. Severe renal dysfunction: estimated creatinine clearance of < 20 mL/min, measured in 24 hour urine or calculated using the formula of Cockroft and Gault
23. History or presence of clinically relevant CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. History of CNS leukemia that is controlled at relapse may be enrolled in this study.
24. History of malignancy other than ALL within 5 years prior to start of protocol-specified therapy with the exception of:

    * Malignancy treated with curative intent and with no known active disease present for 2 years before enrollment and felt to be at low risk for recurrence by the treating physician including
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated cervical carcinoma in situ without evidence of disease
    * Adequately treated breast ductal carcinoma in situ without evidence of disease
    * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
25. Current autoimmune disease or history of autoimmune disease with potential CNS involvement
26. Live vaccination within 2 weeks before the start of study treatment
27. Known hypersensitivity to immunoglobulins or to any other component of the study drug formulation
28. Subject has known sensitivity to immunoglobulins or any of the products or components to be administered during dosing.
29. Currently receiving treatment in another investigational device or drug study or less than 30 days since ending treatment on another investigational device or drug study(s). Thirty days is calculated from day 1 of protocol-specified therapy
30. Subject likely to not be available to complete all protocol-required study visits or procedures, including follow-up visits, and/or to comply with all required study procedures to the best of the subject's and Investigator's knowledge.
31. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
32. Woman of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they fulfil at least one of the following criteria:

    * Post-menopausal (i.e. 12 months of natural amenorrhea or 6 months of amenorrhea with Serum FSH > 40 U/ml
    * Post-operative after bilateral ovariectomy with or without hysterectomy
    * Continuous and correct application of a contraception method with a Pearl index of < 1% (e.g. implants, depots, oral contraceptives, intrauterine device) from initial study drug administration until at least 3 months after the last dose of study drug. A hormonal contraception method must always be combined with a barrier method (e.g. condom)
    * Sexual abstinence
    * Vasectomy of the sexual partner
33. Male who has a female partner of childbearing potential, and is not willing to use 2 highly effective forms of contraception while receiving protocol-specified therapy and for at least an additional 3 months after the last dose of protocol-specified therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Phase I/ part 1: Maximum tolerated dose (MTD) | through study part I completion, anticipated after 1 year
  The primary endpoint of the part I dose escalation part will be maximum tolerated dose (MTD).
  The combination of Venetoclax and Blinatumomab will be evaluated for tolerability in a 3+3 design. In a 3+3 design, three patients will form a cohort. Each cohort will receive a higher cumulative dose of Venetoclax in pre-defined dose escalation steps (see table below). If one patient experiences dose limiting toxicity (DLT), the cohort will be expanded to six patients.
  If two or more of these 6 patients experience a DLT, the next lower Venetoclax dose will be defined as maximum tolerated dose (MTD). If 0/3 or <2/6 patients in a cohort experience a DLT, the next dose escalation cohort will be opened. In case of ≥ 2 DLTs at the dose level 1, dose level -1 will be used as a fallback option. The DLT evaluation period is defined as the first 49 days after initiation of Venetoclax in cycle 1 (i.e. C1D-7 to C1D42)
Phase II/ part 2: rate of complete molecular remissions (Mol-CR) | after one cycle of treatment (up to 43 days)
  The primary efficacy measure of the part II expansion part will be the rate of complete molecular remissions (Mol-CR) after one cycle of Blinatumomab and Venetoclax.
  - Mol-CR is defined as MRD negativity with a sensitivity of at least 10E-04 Disease status will be assessed by bone marrow and peripheral blood analysis at the end of Cycle 1. Bone marrow aspiration is required at any time on study in case peripheral blood analysis is suspicious for progression of disease.

SECONDARY OUTCOMES:
Rate of composite complete remissions (cCR) | until End of Follow-Up (up to 6 months after EOT)
  rate of composite complete remissions (cCR) including CR without complete hematologic regeneration (CRh) and CR with incomplete recovery of peripheral blood counts (CRi) after one treatment cycle
  * CR is defined as having ≤ 5% blasts in the bone marrow, no evidence of disease, and full recovery of peripheral blood counts (i.e. platelets ≥ 100.000/μl, and ANC
    ≥ 1.000/μl), and no evidence of (extramedullary) disease
  * CRh is defined as having ≤ 5% blasts in the bone marrow, no evidence of disease, and partial recovery of peripheral blood counts (i.e. 50.000/μl < platelets < 100.000/μl, and 500/μl < ANC < 1.000/μl), and no evidence of (extramedullary) disease
  * CRi is defined as having ≤ 5% blasts in the bone marrow, no evidence of disease and incomplete recovery of peripheral blood counts (i.e. platelets ≥ 50.000/μl or ANC ≥ 1.000/μl, and no evidence of (extramedullary) disease
Overall response rate (ORR) | until End of Follow-Up (up to 6 months after EOT)
  overall response rate (ORR), including rate of CR, CRh, CRi, and rate of partial remission (PR)
Remission duration | at 1 year and 2 years after EOT
  median and probability of Remission duration at 1 year and 2 years
Event-free survival (EFS) | at 1 year and 2 years after EOT
  o EFS time will be calculated from the time of starting on-protocol therapy (C1D-7) until the date of (a) disease assessment indicating relapse after having achieved CR/CRh/CRi or (b) disease assessment indicating refractory disease after one or two cylces or (c) death, whichever occurs first. All subjects failing to achieve CR/CRh/CRi after the first cycle will be reassessed after two cycles if applicable.
  Subjects alive and relapse-free at the time of analysis will be censored on their last disease assessment date.
Overall survival (OS) | at 1 year and 2 years after EOT
  median OS times will be calculated from the time of starting on-protocol therapy (C1D-7) until death due to any cause. Subjects still alive at the time of analysis will be censored at the date last known to be alive.
Overall response rate (ORR) | after one cycle of treatment (up to 43 days)
  including CR, CRh, CRi and partial remission (PR)
  o PR is defined as having 5% < blasts < 20% in the bone marrow, no evidence of disease, and partial recovery of peripheral blood counts (i.e. platelets > 50.000/μl, and ANC > 500/μl)
CR rates in comparson to Blinatumomab monotherapy | after one cycle of treatment (up to 43 days)
  CR rates in comparson with historical cohorts treated with Blinatumomab alone with inverse probability of treatment weighting (IPTW) using the propensity score
Duration of MRD response | until End of Follow-Up (up to 6 months after EOT)
  Probability of continuous MRD response and complete MRD response and duration of MRD response
Measurement of Quality of Life | until End of Follow-Up (up to 6 months after EOT)
  Measurement of Quality of Life with EORTC instruments (EORTC QLQ C30 and EQ-5D) at different time-points during treatment
Rate of allogeneic stem cell transplantation | until End of Follow-Up (up to 6 months after EOT)
  Proportion of patients who undergo allogeneic stem cell transplantation
Relapse localisations | until End of Follow-Up (up to 6 months after EOT)
  Frequency of different relapse localisations in proportion to total hematological relapses

OTHER OUTCOMES:
Treatment realisation 1 | until end of treatment (up to 1+12 weeks)
  incidence of treatment interruptions
Treatment realisation 2 | until end of treatment (up to 1+12 weeks)
  total dose reductions
Treatment realisation 3 | until end of treatment (up to 1+12 weeks)
  total treatment discontinuations

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Goekbuget, MD, Principal Investigator — GMALL-Study-Group
Locations (17):
- Germany (17):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - University Hospital of Frankfurt (Main), Frankfurt am Main, Hesse
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Charité - Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Köln, Cologne
  - University Hospital Düsseldorf, Düsseldorf
  - Universität Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - UKSH-Kiel, Kiel
  - Universitätsklinik Leipzig, Leipzig
  - Klinikum Mannheim, Mannheim
  - Klinikum Rechts der Isar der TU München, München
  - Klinikum Oldenburg, Oldenburg
  - Robert - Bosch - Krankenhaus, Stuttgart

IPD SHARING:
Plan to Share IPD: No